CLINICAL TRIAL: NCT04807647
Title: The Effect of White Noise on Sucking Success and Baby Comfort in Premature Babies
Brief Title: the Effect of White Noise on Sucking and Baby Comfort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Esra Tanrıverdi (Other)
Responsible Party: Sponsor-Investigator, Esra Tanrıverdi, Research Assistant, Zonguldak Bulent Ecevit University
Organization: Zonguldak Bulent Ecevit University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 12102020100153
Record Dates: First submitted 2021-02-17; First posted 2021-03-19 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Sucking Behavior
Keywords: newborn; music; comfort
MeSH Terms: conditions — Sucking Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music band (Experimental): The starting person will first talk about white noise and explain how he can direct breastfeeding, and fill the Informed Volunteer Form, Patient Identification Form and Application Registration Form. The mother and baby will be given the appropriate position and breastfeeding will be started. No application will be applied to the mother during the first breastfeeding. During the second breastfeeding, 30 newborn group Orhan OSMAN's "Kolik" album will be played on the music player "Your Baby Don't Cry". After the process is completed, a written response will be received for the data Premature Baby Comfort Scale, LATCH breastfeeding diagnostic measurement tool, Patient Diagnosis Form and Application Registration Form.
  Interventions: Other: Orhan OSMAN's track "Don't Let Your Baby Cry" in the "Kolik" album will be played on the music player.
- control (No Intervention): First, the mother will be informed about the study. Then the appropriate position will be given. The informed volunteer form, the Patient Identification Form and the Application Registration Form will be filled. The mother and the baby will be given the appropriate position and breastfeeding will be started. No application will be applied to the mother during the first breastfeeding. No intervention will be applied during the second breastfeeding. After the procedure is completed, a written response will be received with the data Premature Infant Comfort Scale, LATCH breastfeeding diagnostic measurement tool, Patient Diagnosis Form and Application Registration Form.

INTERVENTIONS:
Other: Orhan OSMAN's track "Don't Let Your Baby Cry" in the "Kolik" album will be played on the music player. — white noise will be played while breastfeeding
  Arms: music band

SUMMARY:
The study is a randomized controlled study to determine the effect of white noise on sucking success and infant comfort in newborns in babies aged 34-37 weeks who were fed orally by a full enteral mother in the Neonatal Intensive Care Unit.

DETAILED DESCRIPTION:
The Type and Purpose of the Research

The study is a randomized controlled study to determine the effect of white noise on sucking success and infant comfort in newborn babies between 34-37 weeks of gestation who were fed orally by a full enteral mother hospitalized in the Neonatal Intensive Care Unit.

Place and Time of the Study

The research was conducted in the Bulent Ecevit Training and Research Hospital Neonatal Intensive Care Unit between 01.09.2020 and 01.03.2021.

MATERIAL AND METHOD OF THE RESEARCH

The study is a randomized controlled study to determine the effect of white noise on sucking success and infant comfort in newborn babies between 34-37 weeks of gestation who were fed orally by a full enteral mother hospitalized in the Neonatal Intensive Care Unit.

Research Universe

The universe of the study consisted of newborn babies who were born in the Bulent Ecevit Training and Research Hospital Neonatal Intensive Care Unit between 01.09.2020 and 01.03.2021 and who met the inclusion criteria in the study and the babies who were fed by the mother who passed to the mother's room.

Research Sample Thirty control newborn infants who volunteered to participate in the study and met the inclusion criteria were formed by 30 newborns in the white noise group.

Sampling Selection Criteria

* Gestational age between 34-37 weeks,
* Having a birth weight of 1800-3600 g,
* Does not have any anatomical and physiological problems,
* Does not show any signs of disease and does not have any congenital disorder,
* Does not have a congenital or acquired malformation related to hearing
* Families without any disability to breastfeed
* Having parental consent

Materials and Methods

In this study, babies who were called to feed mothers who started to be fed orally with breast milk after leaving intensive care were selected. Informed consent form, Patient Identification Form and Application Registration Form, Premature Infant Comfort Scale, and LATCH Breastfeeding Diagnostic Measurement Tool were used for parents who accepted to participate in the study. The control group and the intervention group were first told about white noise and how it could affect breastfeeding, and the Informed Volunteer form, the Patient Identification Form and the Application Registration Form were filled. The mother and the baby were given the appropriate position and breastfeeding was initiated. No application was applied to the mother during the first breastfeeding. During the second breastfeeding, 30 neonatal groups were listened to the song "Your Baby Don't Cry" from Orhan OSMAN's album "Kolik". During the second breastfeeding, no music was played to the control group. After the procedure was completed, the data were collected by the researcher using the Premature Baby Comfort Scale, LATCH breastfeeding diagnostic measurement tool, Patient Diagnosis Form and Application Registration Form. Then the data will be analyzed in the spss 16.0 package program.

Data Collection Tools

* Introductory Information Form for Mother and Baby
* LATCH Breastfeeding Diagnostic Scale
* Premature Baby Comfort Scale Decibel measuring device
* Orhan Osman's Colic album-Don't Let Your Baby Cry II

ELIGIBILITY:
Inclusion Criteria:• Gestational age between 34-37 weeks,

* Having a birth weight of 1800-3600 g,
* Does not have any anatomical and physiological problems,
* Does not show any signs of disease and does not have any congenital disorder,
* Does not have a congenital or acquired malformation related to hearing
* Families without any disability to breastfeed
* Having parental consent

Exclusion Criteria:

* • Gestational age cannot be between 34-37 weeks

  * Birth weight not in the range of 1800-3600,
  * Having any anatomical and physiological problems
  * Any signs of illness and congenital disorder
  * Having a congenital or acquired malformation related to hearing
  * Families who have any disability to breastfeed
  * No parental consent

Ages: 34 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
LATCH Breastfeeding Diagnostic Measurement Tool | 2-6 month
  This measurement tool consists of five evaluation items, a combination of the first letters of these items. The item is between 0 and 2 points. The highest score that can be obtained from the scale is ten. The measurement tool does not have a cut-off point and the higher the LATCH score, the better the breastfeeding success is evaluated.If we look at the five criteria, breast retention, Seeing the swallowing movement of the baby, Type of nipple, Comfort of dyeing the mother's breast and nipple, Holding the baby is the position.

SECONDARY OUTCOMES:
Premature comfort scale | 2-6 month
  It was developed to measure the pain and stress levels of 0-18 years old children hospitalized in the intensive care unit.
  It is considered as 7 parameters such as Physical Movement, Muscle Tone, Facial Movements and Average Heart Rate. Each group is a 5-point Likert type scored from 1 to 5, from bad to good. Accordingly, the comfort of the baby is interpreted on the total score. According to this score, 35 is the lowest and 7 the highest comfort score. A high score on the scale indicates that the baby's comfort level is low. If the total score received is 17, the cut-off value of the scale is the limit for the baby's comfort level, indicating the need for an intervention to reduce pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit Eğitim Araştırma Research Hospital, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study protocol